CLINICAL TRIAL: NCT02215889
Title: A Phase I/II Clinical Trial to Evaluate the Benefit and Efficacy of Liver Resection And Partial Liver Segment 2/3 Transplantation With Delayed Total Hepatectomy as Treatment for Selected Patients With Liver Metastases From ColoRectal Carcinoma
Brief Title: Partial Liver Segment 2/3 Transplantation Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Smedman, MD, M.D, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAPID 2014
Record Dates: First submitted 2014-06-24; First posted 2014-08-13 (Estimated); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: Liver metastases; Transplantation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental)
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation

SUMMARY:
The patients will receive hepatectomy as a 2 stage procedure. In the first surgical procedure liver segments 2-3 are removed and liver donor segments 2-3 inserted. After growth of donor segments 2-3, the remaining liver segments of the recipient are removed. The patient will at this time have only donor liver tissue in place.

ELIGIBILITY:
Inclusion Criteria:

* Histologically verified adenocarcinoma in colon/rectum.
* Liver metastases, not amenable to liver resection
* No signs of extra hepatic metastatic disease or local recurrence according to PET/CT scan within 4 weeks prior to the faculty meeting at the transplant unit, except patients may have 1-3 resectable lung lesions all<15mm.
* No signs of extra hepatic metastatic disease on CT thorax/abdomen/pelvis within 4 weeks prior to the faculty meeting at the transplant unit, except patients may have 1-3 resectable lung lesions all<15mm.
* No local recurrence according to MR-pelvis scan in patients with rectal cancer within 4 weeks prior to the faculty meeting at the transplant unit
* No signs of local recurrence judged by colonoscopy / CT colography within 12 months prior to the faculty meeting at the transplant unit
* Good performance status, ECOG 0 or 1.
* Satisfactory blood tests: Hb >10g/dl, neutrophiles >1.0 (after any G-CSF), TRC >75, Bilirubin<2 x upper normal level, ASAT,ALAT<5 x upper normal level, Creatinine <1.25 x upper normal level. Albumin above lower normal level.
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to GCP, and national/local regulations.
* All patients should have received at least 8 weeks of chemotherapy.

Exclusion Criteria:

* Weight loss >10% the last 6 months
* Patient BMI > 30
* Previous diagnosed bone or CNS metastatic disease.
* Previous diagnosed cancer mammae or malignant melanoma.
* Palliative resection of primary CRC tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2025-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Percent of transplanted patients receiving second stage hepatectomy within 4 weeks of segment 2/3 transplantation. | 4 weeks

SECONDARY OUTCOMES:
Overall Survival | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Norway